CLINICAL TRIAL: NCT03074903
Title: Does Skyla Insertion Timing Impact Bleeding?
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Noaa Shimoni, Assistant Professor, Family Medicine, NJMS, Rutgers, The State University of New Jersey
Other Study IDs: Pro20150001449
Record Dates: First submitted 2017-02-06; First posted 2017-03-09 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Vaginal Bleeding
Keywords: intrauterine device; bleeding
MeSH Terms: conditions — Uterine Hemorrhage; Hemorrhage | interventions — Intrauterine Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Early cycle insertion: Participants in this group have the intrauterine system inserted during the first seven days of their menstrual cycle.
  Interventions: Device: Intrauterine system
- Late cycle insertion: Participants in this group have the intrauterine system inserted during the remainder of their cycle.
  Interventions: Device: Intrauterine system

INTERVENTIONS:
Device: Intrauterine system — Women having the Skyla intrauterine system at different times during their menstrual cycle report their bleeding patterns through daily texts.
  Other Names: Intrauterine device

SUMMARY:
Women presenting for contraception will be offered the IUS Skyla and study participation. Daily bleeding will be collected for a total of 90 days and correlated with insertion timing and baseline endometrial thickness.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45
* Parous or nulliparous
* Desire Skyla for contraception
* Regular menstrual cycles (21-35 days)
* Working mobile phone and willing to accept text messages and report daily bleeding data for 90 days

Exclusion Criteria:

* Vaginal or cesarean delivery in the past 12 weeks
* Abortion in the past 6 weeks
* Uterine anomaly distorting the uterus
* Acute pelvic inflammatory disease
* Uterine bleeding of unknown etiology
* Acute liver disease or tumor
* History of progestin-sensitive cancer
* Abnormal pap smear awaiting diagnostic or therapeutic intervention

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women presenting for intrauterine device insertion.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2016-04-16 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Bleeding and spotting as collected by daily texts | 90 days
  Composite variable of bleeding and spotting for 90 days after Skyla IUS insertion

CONTACTS AND LOCATIONS:
Overall Officials: Noa'a Shimoni, MD MPH, Principal Investigator — Rutgers University
Locations (3):
- United States (3):
  - Planned Parenthood, Morristown, New Jersey
  - NJFPC, Newark, New Jersey
  - SHS, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimoni N, Choudhury T, Goldman AR, Frondelli M, Chen PH. Bleeding and spotting with the levonorgestrel 13.5 mg intrauterine system: the impact of insertion timing. Contraception. 2019 Jun;99(6):340-344. doi: 10.1016/j.contraception.2019.02.004. Epub 2019 Mar 1. PMID 30831104